CLINICAL TRIAL: NCT03587870
Title: Protein Delivery in Intermittent and Continuous Enteral Nutrition in ICU Patients A Prospective, Randomised Controlled Pilot Study in Critical Ill Patients With a Protein-rich Formula
Brief Title: Protein Delivery in Intermittent and Continuous Enteral Nutrition in ICU Patients
Acronym: ProBoNo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EKNZ 2018-00259
Record Dates: First submitted 2018-06-04; First posted 2018-07-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Muscle Wasting in Critically Ill
Keywords: intensive care unit; intermittent enteral nutrition; continuous enteral nutrition; muscle wasting
MeSH Terms: conditions — Muscular Atrophy | interventions — Enteral Nutrition

STUDY DESIGN:
Intervention Model Description: A prospective, randomised controlled pilot study in critical ill patients with a protein-rich formula
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus enteral nutrition with Fresubin Intensive (Experimental): Bolus nutrition over 30-40 minutes every 4 hours with Fresubin Intensive
  Interventions: Other: Enteral nutrition with Fresubin Intensive
- Continuous enteral nutrition with Fresubin Intensive (Active Comparator): Continuous nutrition over 20 hours per day with Fresubin Intensive (standard)
  Interventions: Other: Enteral nutrition with Fresubin Intensive

INTERVENTIONS:
Other: Enteral nutrition with Fresubin Intensive — Comparison of intermittent (experimental) vs continuous (standard, active comparator) enteral nutrition on muscle wasting in critically ill patients

SUMMARY:
Acute skeletal muscle wasting in ICU patients is associated with functional impairment and with increased risk of death. Of what we know today, physical disability can persist up to 5 years. Adequate nutrition is the basis for an optimal recovery for ICU patients and for prevention of muscle wasting. Today, continuous feeding is still the standard enteral nutrition form for patients in the ICU to limit the incidence of aspiration. A study of Serpa et al. and Georgia et al. compared the continuous feeding versus a bolus nutrition with a feeding time of 30 - 60 minutes every 4 hours. They showed no statistical differences in complications between both groups.

ProBoNo is a prospective, randomized, controlled pilot study of critically ill patients with a protein- rich formula to explore the impact of continuous or intermittent bolus nutrition on muscle breakdown in ICU patients. The investigators would like to recruit 68 patients during the first 24 hours after surgical intensive care unit admission. Prior beginning of nutrition administration, and on the 7th day thereafter the investigators will perform a muscle biopsy and an ultrasound from the vastus lateralis muscle in both groups.

The primary outcome is the time from 6.00 am of the following day after admission until the patient reaches his daily protein's target quantity. Secondary outcomes include the diameter and densitiy of the hamstrings assessed by ultrasound and histology, the process of gastric residual volume, number of diarrhoea events and laboratory findings like glucose, urea and insulin like growth factor (IGF)-1, all compared between the two time points.

Intermittent feeding is not only more natural and could help to limit the muscle wasting in ICU patients, it is also easier to handle for the ICU caring medical team. A trial from Georgia et al. in 2007 compared continuous to intermittent enteral nutrition. They found that the intermittently fed patients reached their nutrition goal faster than those being continuously nourished. This might in part be explained by feeding interruptions in the continuous feeding regimen. Presumably, preoperative holding of tube feedings in the continuous nutrition group most commonly caused interruptions. Thus, independently from prevention of muscle breakdown, a bolus nutrition would be more attractive.

DETAILED DESCRIPTION:
The relevance of early continuous or intermittent enteral feeding of critically ill patients has been discussed controversially in the last years. Today, continuous feeding is still the standard for enteral nutrition in the ICU. The continuous nutrition can prevent abdominal intolerance like vomiting, diarrhoea and aspiration. Pulmonary aspiration is the most dramatic consequence of enteral nutrition and can be limited by a continuous feeding as shown by a study in 2003. However, nutrition was started with a bolus of 125ml as baseline by force of gravity over 15 minutes. Compared to the continuous nutrition, this is considered much volume in a short time. Naturally, risk of gastric intolerance in this scenario is very high.

In other studies, a similar amount of nutrition was given over a longer period of time (30 - 60 minutes) every 4 hours. In each cohort (continuous and bolus), only one case of pulmonary aspiration or tube obstruction was detected. After this study, other trials with a similar result followed. In 2007 a trial of Georgia et al. showed no statistical differences in complications regarding tube feeding, no differences of diarrhoea, emesis or pneumonias between continuous and bolus nutrition. The feeding time for bolus nutrition is also a critical influential factor. When an intermittent feeding is given over a longer period of time (20-40 minutes), the incidence of nausea and vomiting has not increased.

Intermittent feeding is not only a good alternative to continuous feeding, but also more natural, as long-term intake of nutrition over 20 hours is not common in any mammal. The alimentary tract and metabolic pathways of humans seem designed for intermittent ingestion of essential nutrients reduced to a few times a day. Different hormones of the endocrine cells affect complex roles of gastrointestinal motility, gall bladder contraction and nutrient absorption. The level of these hormones depends on the amount of nutrient ingestion. This response of the hormones is almost completely abolished in continuous feeding. But in intermittent nutrition, hormones like incretin, glucose-dependent insulinotropic polypeptide (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP) boost the level of insulin and the resulting carbohydrate load and therefore influence the muscle protein synthesis and breakdown.

In healthy individuals, the anabolic effects of feeding occur due to an increase on the synthetic rate of muscle protein synthesis of approximately 300% with a simultaneous 50% decrease in the rate of protein breakdown. Two studies of 2009 and 2011 compared the intermittent bolus and continuous feeding and the effect of protein synthesis in skeletal muscle in neonatal pigs. They analysed the fractional rates of protein synthesis in muscle samples of continuous and intermittent bolus feeding groups. They could show that although both groups, continuous and intermittent bolus feeding, stimulate muscle protein synthesis, but in the bolus-fed, in the fractional rates of protein synthesis called K's was greater after a meal.

An ongoing study wants to show the effect of bolus vs. continuous feeding in ICU patients related to muscle wasting by measurements of ultrasound and blood samples. In this trial, the investigators would like to have a similar approach but with different measurements. Using ultrasound and muscle biopsies, the investigators aim to determine whether intermittent enteral feeding could preserve muscle mass better or more than standard continuous enteral feeding in the critically ill patients. In addition, the investigators would like to assess if intermittent bolus feeding optimizes protein intake in the first 7 days of critical illness since the intermittent route is less affected by interruptions following treatment and diagnostic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Adult patients (age 18 years or older)
* Expected ICU stay of five days or longer
* Expected enteral feeding during at least five days

Exclusion Criteria:

* Pregnancy or breast feeding (women of childbearing age are tested for high beta-human chorionic gonadotropin (hCG) in urine or serum upon ICU admission)
* Clinically significant chronic or acute kidney insufficiency with a glomerular filtration rate (GFR) <15.
* BMI ≤ 18 and ≥ 35.
* Intestinal perforation, peritonitis, intestinal fistula, necrosis or other contraindication to enteral diet
* Death or discharge before 48 hours of observation
* Noradrenaline ≥ 0.5 µg/kg bodyweight /min
* Inherited and chronic skeletal muscle disease (e.g. Morbus Duchenne or other motoneuron disease)
* Paralysis (e.g. hemiplegia, tetraplegia and paraplegia)
* Immunosuppression
* Haematologic malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Daily protein target quantity | During ICU stay for the duration of 7 days after study inclusion
  Is the time from 6.00 am of the following day after admission until the patient reaches his daily protein target quantity (1.2 g/ kg Biologische Wertigkeit (BW)/ biological value protein in the control group, to 1.5 g/kg BW protein in the experimental group).

SECONDARY OUTCOMES:
Diameter of the hamstrings | During ICU stay, exactly 7 days after study inclusion
  Diameter of the hamstrings assessed by ultrasound and histology
Gastric residual content | Every day during ICU stay for the duration of 7 days after study inclusion
  Amount of gastric residual volume (ml)
Diarrhoea | Every day during ICU stay for the duration of 7 days after study inclusion
  Number of diarrhoea events
Glucose (mmol/l) measurement | Every day during ICU stay for the duration of 7 days after study inclusion
  Laboratory parameters relevant to assess under enteral Nutrition (Glucose (mmol/l))
BUN (mg/dl) measurement | Every day during ICU stay for the duration of 7 days after study inclusion
  Laboratory parameters relevant to assess under enteral Nutrition (BUN (mg/dl))
IGF-1 (mmol/l) measurement | Every day during ICU stay for the duration of 7 days after study inclusion
  Laboratory parameters relevant to assess under enteral Nutrition (IGF-1 (mmol/l))

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Hollinger, MD, Principal Investigator — University Hospital Basel, Basel Switzerland
Locations (1):
- University Hospital Basel, operative ICU, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Reinhold S, Yeginsoy D, Hollinger A, Todorov A, Tintignac L, Sinnreich M, Kiss C, Gebhard CE, Kovacs B, Gysi B, Imwinkelried L, Siegemund M. Protein delivery in intermittent and continuous enteral nutrition with a protein-rich formula in critically ill patients-a protocol for the prospective randomized controlled proof-of-concept Protein Bolus Nutrition (Pro BoNo) study. Trials. 2020 Aug 25;21(1):740. doi: 10.1186/s13063-020-04635-1. PMID 32843075